CLINICAL TRIAL: NCT01888419
Title: A Prospective, Randomized Study of the Possible Pain Relieving and Scar Tissue Modifying Properties of Lipotransplantation in a "Post Breast Therapy Pain Syndrome" Setting
Brief Title: Investigation of the Pain Relieving Properties of Lipotransplantation After Treatment for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Alexander Juhl Andersen, M.D., Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBTPS 1-10-72-76-13
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Pain
Keywords: Post Breast Therapy Pain Syndrome; Lipotransplantation; Breast Cancer; Pain
MeSH Terms: conditions — Chronic Pain; Breast Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No active treatment (No Intervention): Clinical follow-up, no active intervention.
- Lipotransplantation (Experimental): Lipotransplantation in general anaesthesia to the mastectomy site.
  Interventions: Other: Lipotransplantation

INTERVENTIONS:
Other: Lipotransplantation — Lipotransplantation in general anaesthesia to the mastectomy site
  Other Names: Fat grafting; Fat transplantation
  Arms: Lipotransplantation

SUMMARY:
Background

In Denmark, breast cancer is the most common fatal cancer in women with more than 4700 new cases annually. Unfortunately, up to 60% of women who are treated surgically for breast cancer, will experience chronic pain as a consequence of the treatment. This state of chronic neuropathic pain is termed "Post Breast Therapy Pain Syndrome" or PBTPS.

The purpose of the study

The purpose of this study is to investigate whether transplantation of fat cells (lipotransplantation) to the pain affected mastectomy area, could have an analgesic effect in women who have developed PBTPS. Secondary, we wish to investigate if lipotransplantation has a beneficial effect on the quality of the skin and the scar in the area where the transplanted fat cells are placed.

Hypotheses

* Lipotransplantation to the area under the scar tissue and the area under the pain-afflicted area reduces the pain in women with PBTPS.
* The neuropathic pain in PBTPS is correlated to the number of free nerve endings crossing the border between the dermis and the epidermis
* Lipotransplantation have a beneficial effect on the scar tissue structure and improves the skin quality.

Patients

Women who have undergone treatment for breast cancer and subsequently developed PBTPS. A total of 32 patients with PBTPS will be included.

Methods

Patients will be randomly assigned to receive either lipotransplantation or no active treatment. At three follow-up visits, the perceived pain of the patient and the skin and scar quality will be scored. In addition, a 3-mm biopsy will be taken from the skin on both the missing and the healthy breast, and from the mastectomy scar.

The scoring of the perceived pain and the quality of the skin and the scar, allows us to investigate if the lipotransplantation have an effect on pain, and skin/scar quality. Additionally, the skin and scar biopsies will be examined on a microscopic level, in order to investigate why lipotransplantation has these effects.

Conclusion

In summary, the results of this project could help to increase our understanding of why some patients develop chronic neuropathic pain after mastectomy and radiotherapy. It is our hope that our results may contribute to the development of better and more effective treatment that will be beneficial for the project participants and future patients.

DETAILED DESCRIPTION:
Background

In Denmark, breast cancer is the most common fatal cancer in women with more than 4700 new cases annually. All patients are treated according to national guidelines developed by the Danish Breast Cancer Cooperative Group (DBCG). Treatment primarily consists of surgical removal of all or parts of the breast and simultaneous removal of one-or lymph nodes in the ipsilateral axilla. Subsequently, there may be a need for additional treatment with chemotherapy, radiation and / or anti-hormonal therapy, in order to reduce the risk of recurrence.

Up to 60% of women who are treated surgically for breast cancer, will experience chronic pain as a consequence of the treatment. This condition was previously referred to as "Post Mastectomy Pain Syndrome", but because the condition is also seen after less extensive forms of breast cancer surgery, the condition is now termed "Post Therapy Breast Pain Syndrome" (PBTPS). PBTPS is defined as a neuropathic pain condition with pain localized to the axilla, the medial part of the upper arm, chest and or chest wall of the side of surgery, lasting more than three months after surgery and / or the end of treatment.

In 2011 Caviggioli et al. published a study where lipotransplantation to the mastectomy area was found to have a significant analgesic effect. The aforementioned study is to date the only published study in the field. However, it is not a randomized study. In order to obtain further evidence of the apparent beneficial effect of lipotransplantation on pain, the present study has been initiated.

Lipotransplantation is a fast and relatively non-invasive technique which is described in detail by Coleman et al.. Additionally, in a study from 2008, Klinger et al. found that lipotransplantation to burn scars in the face resulted in a significant improvement in the patient's skin and scar quality and also reduced pain in the treated areas. The theoretical basis for the scar and skin modifying effects of lipotransplantation has not yet been finally understood. To the best of our knowledge, no studies have systematically investigated and analysed the effects of lipotransplantation on the irradiated mastectomy area on a histological level.

The purpose of the study

The purpose of this study is to investigate whether lipotransplantation to the pain affected mastectomy area, could have an analgesic effect in women affected by Post Breast Therapy Pain Syndrome. Secondary, we wish to investigate the scar and skin modulating effects of lipotransplantation to the same area.

By carrying out immunohistochemical staining and subsequent stereoscopic microscopy of free nerve endings in the skin biopsies taken before and after lipotransplantationen we wish to determine whether changes in the number and type of free nerve endings is part of the mechanism of pain reduction.

Hypotheses

* Lipotransplantation to the area under the scar tissue and the area under the pain-afflicted area reduces the pain in women with PBTPS.
* The neuropathic pain in PBTPS is correlated to the number of free nerve endings crossing the border between the dermis and the epidermis
* Lipotransplantation have a beneficial effect on the scar tissue structure and improves the skin quality.

Patients

Women who have undergone unilateral mastectomy for breast cancer at Aarhus University Hospital, Aarhus, Denmark and, if applicable, has finished their adjuvant postoperative radiation therapy at least 6 months ago. Patients must have had pain localized to the area of the missing breast for at least three months after adjuvant radiation therapy ended. A total of 32 patients with PBTPS will be included.

Methods

Patients with PBTPS are randomly assigned to receive either lipotransplantation or no active treatment.

Regardless of randomization, the patient will be invited to three follow-up visits, respectively 3 and 6 months after inclusion/surgery. At each of the outpatient visits the participant will be asked to complete the DoloTest ® , VAS pain score and the Patient Scar Assessment Scale. The clinician will complete the Observer Scar Assessment Scale and record the consumption of pain medication. DoloTest ® is a validated, visual analogue questionnaire designed to assess the patients experienced pain and impact on the patients daily life. Three 3-mm punch biopsies will be taken at inclusion, one from the mastectomy scar, one from the skin 2 cm above the mastectomy scar in the medioclavicular line, and one from the healthy skin on the health breast in an area corresponding to the other skin biopsy.

The skin punch biopsies from the pain afflicted area will be fixed in 4% phosphate buffered paraformaldehyde. After freezing, the tissue samples are cut into 50-micron thick sections. Systematically sampled sections immunostained with rabbit anti-human Protein Gene Product 9.5 (a neuron-specific protein), and DAB-marked goat anti-rabbit as the secondary antibody. The sections are then microscoped in an Olympus BX51 light microscope with an Olympus DP71 digital camera and Prior motorized board connected to a computer with Newcast stereology software. Two goals can then be calculated: 1) the number of free nerve endings, which crosses the border between dermis and epidermis per mm 2) the average nerve fibre length density in the epidermis and / or dermis.

The skin punch biopsies from the mastectomy scar are fixed in formaldehyde for embedding in paraffin. The tissue samples are cut into 1-2 micron thick sections and stained with Picrosirius red (PR) colour. By using polarized light microscopy, the various subtypes of collagen fibres may be visualized and differentiated. The thicker collagen fibres (type I) are red-orange-yellow and the thinner collagen fibres (type III) are green. Furthermore, the sections will be stained for elastin. Quantitatively, by means of the above-mentioned method, changes in the volume fraction of collagen type I and III, and elastin may be measured.

Statistical analyzes

The minimal clinically relevant difference the study is looking for, is a Visual Analog Pain score difference of 3. The common standard deviation was estimated from a similar study by Caviggioli et al. in 2011, and set to be 2.96 on the Visual Analog Pain scale. We assume that our standard deviation (SD) will be the same. Using the following formula: N = (Za + Zb)2 x SD2 / dif2 where Za and Zb are the standardized normal deviations corresponding to the selected levels of significance, SD is Standard Deviation and dif is the minimal clinically relevant difference the study is looking for. The result is 16 patients in each arm, totalling 32 patients, when the significance level is set at 5% and the power of the study is set to 80%. Statistical analyzes will be performed in collaboration with a biostatistician from the Health Sciences Institution, Aarhus University, Denmark.

Economic Conditions

The project is supported by: Faculty of Health Sciences, University of Aarhus with three full time equivalents, which is used to pay for full-time academic staff. Other project expenses are to be covered by independent foundations and endowments that do not have an influence on the study. None of the personnel in the project have a financial interest in the project.

Compensation to the participating patients

The participating patients in the study will not receive any financial compensation. However, documented travel expenses will be reimbursed.

Recruitment of participants

Patients are primarily recruited from a previous study, were a questionnaire was sent to all women having received an unilateral mastectomy at Aarhus University Hospital, in the period from 2009 to 2013. In the questionnaire, patients were asked to evaluate their pain in the different areas pertaining to PBTPS, and if they would allow our department to contact them in regards to the present study. If patients fulfilled the inclusion criteria, they are contacted by the primary investigator by telephone, and a meeting were the details of the study are presented is arranged. Patients with PBTPS could also be recruited during their routine visits at the department of oncology.

The patients will always be offered at least 24 hours of consideration before deciding to give written consent to participate in the study. With the signing of the consent form, the patient accepts the terms and conditions in the study. The patient may at any time and without justification withdraw her consent to participate, without her decision affecting her present or future treatment or any other rights the patient may have.

Publication of results

Negative, inconclusive and positive results from the study will be published in internationally recognized, peer-reviewed, English-language journals with an interest in the field.

Ethical statement, side effects and risks

In the present project, data will be treated confidentially in accordance with the Danish Act on Processing of Personal Data. Participants shall be informed both in writing and orally prior to deciding to participate in the study. The participants are thus fully aware of the projects purpose, background and methods, as well as what is expected from the patient's role as a participant.

The participating patients are in the lipotransplantation group, offered an active treatment, which if the current study program can confirm the foreign study, hopefully reduces their daily pain and discomfort and thereby also their consumption of analgesia. If the project provides positive results, the control group will, after the study has ended, be offered the same active treatment.

The patients, which only after informed consent, is part of the project will, in connection with:

1. Lipotransplantation in general anaesthesia; only be exposed to the risk associated with general anaesthesia. The patients in the present study have in relation to their previous surgery for breast cancer been exposed to one or more interventions in general anaesthesia.
2. Risks related to the actual lipotransplantation. At the donor site, there is a risk for short-term tenderness and temporary discolouration. In the long term, a slightly rough surface of the skin may arise. The advantage of the harvest of the fat graft is that the patient achieves a visible improvement of the contour at the donor site.
3. The risk related to the skin punch biopsies: apart from a small scar 1-3 mm corresponding to the place where the biopsy is collected, there is not assessed to any risk of permanent injury or damage.

All interventions are carried out by experienced specialists in plastic surgery with several years experience with lipotransplantation. The general anaesthesia is performed by specialists in anaesthesiology, which are all part of the permanent team at the plastic surgery department and therefore familiar with providing anaesthesia during the described procedures.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosed with and finished treatment for breast cancer
* Unilateral mastectomized
* Finished post operative radiotherapy minimum 6 months ago, if applicable.
* Pain in the area around the missing breast for minimum three months after radiotherapy was finished
* Pain equal to or above 3 on the Numeric Rating Scale for pain
* Verbal and written informed consent

Exclusion Criteria:

* Active breast cancer recurrence
* Other cancer disease
* Pain in the region around the removed breast before the mastectomy
* Active smokers
* Psychiatric illness that prevents informed consent
* Not able to understand and speak Danish
* Patients diagnosed with generalized pain conditions

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pain in the mastectomy area | one year
  The pain in the area around the mastectomy will be measured using visual analog scales (DoloTest), at inclusion of the patient, and at three follow-up visits 3, 6 and 12 months after inclusion.

SECONDARY OUTCOMES:
Collagen in the mastectomy scar | One year
  Changes in the proportions of collagen type I and III in the mastectomy scar.
Elastin content in the mastectomy scar | One year
  Changes in the elastin content of the mastectomy scar.
Free nerve endings crossing between the dermis and the epidermis | One year
  Changes in the number of free nerve endings crossing the border between the dermis and the epidermis per millimeter in the skin of the pain afflicted area around the mastectomy scar.
Mastectomy scar quality | One year
  Changes in the mastectomy scar quality, measured using the Patient and Observer Scar Assessment Scale.
Analgesic consumption | One year
  Changes in the analgesic consumption of the patients included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Juhl Andersen, M.D., Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Background] Carpenter JS, Andrykowski MA, Sloan P, Cunningham L, Cordova MJ, Studts JL, McGrath PC, Sloan D, Kenady DE. Postmastectomy/postlumpectomy pain in breast cancer survivors. J Clin Epidemiol. 1998 Dec;51(12):1285-92. doi: 10.1016/s0895-4356(98)00121-8. PMID 10086821
- [Background] Wallace MS, Wallace AM, Lee J, Dobke MK. Pain after breast surgery: a survey of 282 women. Pain. 1996 Aug;66(2-3):195-205. doi: 10.1016/0304-3959(96)03064-3. PMID 8880841
- [Background] Lundstedt D, Gustafsson M, Steineck G, Malmstrom P, Alsadius D, Sundberg A, Wilderang U, Holmberg E, Johansson KA, Karlsson P. Risk factors of developing long-lasting breast pain after breast cancer radiotherapy. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):71-8. doi: 10.1016/j.ijrobp.2011.05.065. Epub 2011 Nov 11. PMID 22079722
- [Background] Macdonald L, Bruce J, Scott NW, Smith WC, Chambers WA. Long-term follow-up of breast cancer survivors with post-mastectomy pain syndrome. Br J Cancer. 2005 Jan 31;92(2):225-30. doi: 10.1038/sj.bjc.6602304. PMID 15655557
- [Background] Peuckmann V, Ekholm O, Rasmussen NK, Groenvold M, Christiansen P, Moller S, Eriksen J, Sjogren P. Chronic pain and other sequelae in long-term breast cancer survivors: nationwide survey in Denmark. Eur J Pain. 2009 May;13(5):478-85. doi: 10.1016/j.ejpain.2008.05.015. Epub 2008 Jul 16. PMID 18635381
- [Background] Vilholm OJ, Cold S, Rasmussen L, Sindrup SH. The postmastectomy pain syndrome: an epidemiological study on the prevalence of chronic pain after surgery for breast cancer. Br J Cancer. 2008 Aug 19;99(4):604-10. doi: 10.1038/sj.bjc.6604534. PMID 18682712
- [Background] Ducic I, Seiboth LA, Iorio ML. Chronic postoperative breast pain: danger zones for nerve injuries. Plast Reconstr Surg. 2011 Jan;127(1):41-46. doi: 10.1097/PRS.0b013e3181f9587f. PMID 21200198
- [Background] Watson PNC, Evans RJ. The postmastectomy pain syndrome and topical capsaicin: a randomized trial. Pain. 1992 Dec;51(3):375-379. doi: 10.1016/0304-3959(92)90223-X. PMID 1491864
- [Background] Eija K, Tiina T, J NP. Amitriptyline effectively relieves neuropathic pain following treatment of breast cancer. Pain. 1996 Feb;64(2):293-302. doi: 10.1016/0304-3959(95)00138-7. PMID 8740607
- [Background] Caviggioli F, Maione L, Forcellini D, Klinger F, Klinger M. Autologous fat graft in postmastectomy pain syndrome. Plast Reconstr Surg. 2011 Aug;128(2):349-352. doi: 10.1097/PRS.0b013e31821e70e7. PMID 21788826
- [Background] Coleman SR, Saboeiro AP. Fat grafting to the breast revisited: safety and efficacy. Plast Reconstr Surg. 2007 Mar;119(3):775-85; discussion 786-7. doi: 10.1097/01.prs.0000252001.59162.c9. PMID 17312477
- [Background] Klinger M, Marazzi M, Vigo D, Torre M. Fat injection for cases of severe burn outcomes: a new perspective of scar remodeling and reduction. Aesthetic Plast Surg. 2008 May;32(3):465-9. doi: 10.1007/s00266-008-9122-1. PMID 18305985
- [Background] Trojahn Kolle SF, Oliveri RS, Glovinski PV, Elberg JJ, Fischer-Nielsen A, Drzewiecki KT. Importance of mesenchymal stem cells in autologous fat grafting: a systematic review of existing studies. J Plast Surg Hand Surg. 2012 Apr;46(2):59-68. doi: 10.3109/2000656X.2012.668326. PMID 22471250
- [Background] Kristiansen K, Lyngholm-Kjaerby P, Moe C. Introduction and Validation of DoloTest((R)): a new health-related quality of life tool used in pain patients. Pain Pract. 2010 Sep-Oct;10(5):396-403. doi: 10.1111/j.1533-2500.2010.00366.x. PMID 20384966
- See also: The Danish Cancer Society: Incidence of breast cancer in Denmark — http://www.cancer.dk/Hjaelp+viden/kraeftformer/kraeftsygdomme/brystkraeft/statistik+brystkraeft/
- See also: The Danish Breast Cancer Group: Responsible for developing national guidelines for the treatment of breast cancer in Denmark — http://www.dbcg.dk